CLINICAL TRIAL: NCT06260787
Title: The Relationship Between Clinical Profiles And The Success Rate Of In Vitro Fertilization Patients - Experience From Indonesia
Brief Title: Clinical Profiles And In Vitro Fertilization Success
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: OBGY-202401.01
Record Dates: First submitted 2024-01-23; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: in Vitro Fertilisation
MeSH Terms: interventions — Fertilization in Vitro

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In Vitro Fertilisation: Patients undergoing in vitro fertilisation at our tertiary fertility center facility
  Interventions: Procedure: In Vitro Fertilisation

INTERVENTIONS:
Procedure: In Vitro Fertilisation — Assisted reproductive technology in the form of in vitro fertilisation

SUMMARY:
This research was carried out to determine if the IVF patients' clinical profile were connected with how successful in their getting pregnant. This was a cross-sectional study which recruited all patients, performed at a major fertility clinic in Indonesia. Our data collection period spanned between January 2017 and December 2021.

DETAILED DESCRIPTION:
This study was conducted to determine whether there is an association between the clinical profile of in vitro fertilization patients and the success of pregnancy after in vitro fertilization in infertility patients.

The research was a cross sectional study using total sampling method, conducted on 223 infertility patients who performed in vitro fertilization at a tertiary fertility center in Bandung, Indonesia within the period January 2017-December 2021. Secondary data using medical records was taken.

We aimed to identify associations between the patient's age, the male partner's age, infertility duration, IVF protocol, fresh/frozen embryo, various infertility etiologies and the pregnancy rate in IVF programs. A p-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* medical record data for in vitro fertilization patients at our facility from January 1,2017 to December 31, 2021

Exclusion Criteria:

* incomplete patient medical record data.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In vitro fertilisation patients undergoing treatment at our facility
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 5 years
  Total number of patients getting pregnant divided by the number of total patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Hanom H Syam, M.D., Ph.D, Principal Investigator — Permanent Staff at the Department of Obstetrics and Gynecology, Universitas Padjadjaran
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Universitas Padjadjaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Anonymised patient data may be requested to the sponsor/primary researcher if required